CLINICAL TRIAL: NCT04905381
Title: Can a Scalable Parenting Program Improve Children's Readiness for School? An Evaluation of the LENA Start Program
Brief Title: Can the Language Environment Analysis Start Program Improve Children's Readiness for School? LENA Program Evaluation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: William Marsh Rice University (Other)
Collaborators: Alief Independent School District (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-8
Record Dates: First submitted 2020-08-05; First posted 2021-05-27 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Language Development

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): Behavioral: This arm receives usual care (control group). This group will attend their usual Alief group sessions.
  Interventions: Behavioral: Usual care
- LENA Star program (Experimental): Behavioral:LENA Star program. Participants who are selected via the lottery to participate in the LENA Star program will complete ten weekly, 1-hour sessions.
  Interventions: Behavioral: LENA Star Program sessions

INTERVENTIONS:
Behavioral: Usual care — This arm receives usual care (control group)
  Arms: Usual care
Behavioral: LENA Star Program sessions — LENA Start is an evidence-based community program designed to engage families and help them learn how to increase conversation with their children during the first few years of life.
  Arms: LENA Star program

SUMMARY:
The objective of the project is to implement the LENA Start Program at the Alief The objective of the project is to implement the LENA Start Program at the Alief Independent School District in Houston, Texas. The purpose of the study is to learn how maternal expectations about language development influence the child's language development. Also, the study will evaluate how much the mothers believe can affect their child's language development. More specifically, the program implementation will serve as a model that other school districts can readily replicate.

DETAILED DESCRIPTION:
The procedures for this study are broken down into four sections. First, we explain how the LENA Start program lottery will randomly assign participants to the control or treatment group. Next, we explain the LENA Start program that the randomly selected study participants will attend. Then, we explain how the LENA system will be used to measure the child's language environment. Finally, we explain the two meetings parents will attend before and after participation in the LENA Start program as part of the evaluation study, including the instruments used for baseline and endline data collection at these meetings.

1. LENA Start program lottery:

   Participants who consent to participate in the LENA Start program lottery will be randomly assigned to either the control group or the treatment group. Only the treatment group will complete the LENA Start program. The control group will complete only the pre-program and post-program surveys.
2. LENA Start Program:

   If a participant joins the study, they will be invited to participate in the LENA Start Program conditionally upon being randomly assigned to the treatment group. In this program, they will meet other parents who have children of the same age, and they will have the chance to learn and discuss important information about their child's language development. The participants will practice tips about how they can put this information into practice with their own child, thereby enhancing their baby's language development and helping him or her be pre-K ready. Each session will last approximately one hour and there will be ten sessions (one per week). Participants will have the chance to choose a time that best suits their schedule and, if they miss a session, they can always arrange a make-up session with the coordinator. The sessions will take place either online through weekly Zoom meetings with the Alief ISD family liaisons or in person at the Alief ISD intermediate campus family centers.

   After each session, participants will be asked to have their child use the LENA recorder for a day. Once the recording is finished, we will arrange for the participant to turn in the recorder to one of the research assistants on the team. If the sessions are conducted virtually, the parent will be expected to do a contactless exchange by leaving the LENA recorder at a designated location and picking up a new one. If the sessions are in person, the parent will be expected to bring the LENA device to the session each week. From the LENA device recording, we will produce a report that describes the child's language development as well as the quality of the language environment each child is exposed to (as described above). In the Group Sessions, we will teach participants how to read the information from the report and how they can act in simple ways to greatly improve their child's language environment and, in consequence, his or her language development.

   Complete Developmental Snapshot:

   About once a month, we will ask participants to complete the Developmental Snapshot Form. This is a parent-completed evaluation of language skills for infants and toddlers focusing on well-established milestones associated with expressive and receptive language skills. It provides developmental age and percentile ranking information compared to age-matched peers
3. LENA Recordings:

   We measure the quality of the language environment at home by using the LENA System. LENA is an integrated processing and cloud-based software package that enables researchers to collect, manage and analyze multiple recordings of children ages 2 months to 48 months. Each parent will be asked to create 14 LENA recordings, two after the pre-program visit, one after each LENA start session, and two after the post-program visit.

   The research team will download the audio file to the study team computer and transfer to a cloud-based software installed at a server that belongs to the LENA Foundation. The audio file will be processed by the software at the LENA server and will return to the research team four pieces of information:

   Adult Word Count: The Adult Word Count is the number of words a child hears from an adult within a specific period of time: 5 minutes, hourly, daily.

   Child Vocalization Count: A child vocalization is counted when a child's speech of any length is surrounded by greater than 300 milliseconds of silence or other sounds which is not child speech. Conversational Turn (CT) Count: A Conversational Turn occurs when a child vocalizes (initiates) and an adult respond, or an adult speaks (initiates) and a child responds. Each time that happens, one turn is counted.

   Automatic Vocalization Assessment: AVA is an automatic assessment, based on the Adult Word Count, the Child Vocalization Count, and on the Conversational Turn Count. AVA measures a child's expressive language, provides an Estimated Mean Length of Utterance, and estimates the child's language development age. our-by-hour raw counts and age-standardized counts of each one of these five measures of a child's language environment. Once these variables are constructed, the research team will then delete the audio file to prevent any unauthorized use of this file and to reduce the chance of breaches of confidentiality.
4. Evaluation Study:

An interviewer from the Rice research team will meet with the participants before and after their participation in the LENA Start program to conduct baseline and endline data collection. These meetings will be conducted either in person at one of the Alief ISD intermediate schools or virtually through phone calls or Zoom video meetings, depending on the implementation plan decided upon by the school district.

Baseline data collection (visit 1):

At the pre-program baseline visit, parents will be asked to complete the surveys listed below and will be asked to take their first recordings using the LENA device.

Survey questionnaires:

Parent Questionnaire: The parent questionnaire will ask questions about the child's time use to assess the quantity of interaction between adults and the children. We will elicit parental beliefs about the importance of language environment for language development and parental self-efficacy.

Language Development Snapshot (LDS): The snapshot provides parents an estimate of their child's developmental age concerning expressive and receptive language skills. LDS total scores and age estimates are highly correlated with standardized observation-based and parent report language and cognitive assessments, an indication of instrument validity StimQ: We will use the StimQ instrument to measure the child's environment. The StimQ is a 39 point scale for measuring cognitive stimulation in the homes of children ages 12 to 36 months. It is based on a questionnaire that is administered to the child's primary caregiver by trained interviewers in an office setting. StimQ measures only the role of the child's primary caregiver in providing cognitive stimulation for the child. The fact that the StimQ does not require a home observation is an important advantage over other instruments as home visitation would not be practical in this context. Another advantage of the StimQ instrument is that it is rich in collecting information about materials and activities related to parent-child language interaction. The StimQ contains four sections. The first section is the Availability of Learning Materials (ALM) Scale, which consists of a list of toys and games appropriate for children between 12 and 36 months old. The scale is further divided into toys and materials that can be used for symbolic play (e.g., doll or action figure, puppets, housekeeping toys, etc.), for art (e.g., crayons), for fine motor skills (e.g., shape-sorter toys, stacking toys, etc), for language (e.g., set of toy letters), or life-size toys/materials (e.g., tricycle). The second section is the Reading Scale. This scale asks if parents ever read books to the child, the names of the children's books the parents read in the near past, the frequency parents read to the child, and the types of books parents read to the child (books that teach shapes, or letters, or activities, etc.). The third section measures Parental Involvement in the Developmental Advance and contains ten items about teaching to the child. The fourth section measures Parental Verbal Responsivity, and it asks about the nature of parent language interaction with the child.

MacArthur Bates CDI: We will use the MacArthur-Bates Communicative Development Inventories (MB-CDIs) to capture important information about children's developing abilities in early language. The Words & Sentences version is are appropriate for children 16-30 months. It contains a 100-word productive vocabulary checklist and a question about combining words.

Complete two 16-hour recording sessions:

At the pre-program meeting, the research assistant will explain to the parent how to use the LENA recorder and answer any questions the parents may have about it. The parent will also receive a package of materials for conducting the first recording.

If the visit is conducted online, the research assistant will ask the parent how they would like to receive the recording materials package. The parent will be able to choose among the following methods for receiving their recording materials package: a) mail, b) contactless delivery by courier (member of the Rice research team will drop off the package on the family's doorstep) or c) contactless pickup from a designated Alief ISD intermediate school. The parent will also be asked to specify how they would like to return the LENA recording package, either a) mail, b) contactless pickup by courier or c) contactless drop-off at a designated Alief ISD intermediate school.

Endline data collection (visit 2):

At the post-program visit, participants will be asked to complete the same questionnaires as at the pre-program visit (the Parent Survey, the Language Development Snapshot, the StimQ) except MacArthur Bates. The participants will also be asked to complete another two 16-hour recordings using the LENA device. The same options for receiving and returning the LENA recording device will be offered to parents and they will be asked to choose their preferred method.

Fidelity of implementation data collection:

At each of the 10 LENA program sessions, a member of the Rice research team will attend (either virtually or in-person) and collect data about Fidelity of Implementation of the LENA program, including liaison adherence to the material in the session, parental behavior at the session, liaison workload and preparation, as well as other measures of fidelity.

Additionally, at the beginning of every session, a Rice research team member will administer a questionnaire to the liaisons as part of the Fidelity of Implementation data collection.

This data will be collected in both the in-person implementation plan or the virtual implementation plan. If sessions are conducted virtually, a member of the Rice research team will join the weekly Zoom meeting. If sessions are conducted in person, the research team member will attend the weekly meetings in Alief schools.

ELIGIBILITY:
Inclusion Criteria:

Eligible adult participants include parents who meet all the criteria listed below.

1. Must be 18 years old or older.
2. Must have a child between 16 and 30 months old as of September 1, 2022.
3. Must speak English or Spanish as their native language.
4. Must live in the catchment area of Alief Independent School District. Children of the adult participants enrolled in the study are eligible to participate. The children must meet all the criteria below.

1. Must be between 16 and 30 months old as of September 1, 2022 2. Must speak English or Spanish as their native language. 3. Must live in the catchment area of Alief Independent School District.

Exclusion Criteria:

Adult participants will not be eligible for this study if they:

* Are NOT 18 years old or older.
* Do NOT have a child between 16 and 30 months as of September 1, 2022.
* Do NOT speak English or Spanish as their native language.
* Do NOT live in the catchment area of Alief Independent School District.

Children will not be eligible for this study if they:

* Are NOT between 16 and 30 months as of September 1, 2022.
* Do NOT speak English or Spanish as their native language.
* Do NOT live in the catchment area of Alief Independent School District.

Ages: 16 Months to 30 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of the Language Environment: Language Environment Analysis (LENA System) | Measured at 16 to 30 months of age
  The quality of the language environment at home will be measured by using the LENA System. LENA is an integrated processing and cloud-based software package that enables researchers to collect, manage, and analyze multiple recordings of children ages 2 months to 48 months.LENA device estimates adult words spoken to and around the key child, adult-child conversational interactions, child vocalizations, and language from Television and/or electronics
Measurement of the Child's Home Environment | Measured at 16 to 30 months of age
  StimQ Availability of Learning Materials Scale (ALM). The availability of learning materials will be measured by using the StimQ ALM scale. The StimQ is a structured interview. Individual items are summed, and scores range ranges from 0 to 7. Higher scores are correlated with better parental behavior.
Measurement of the Child's Home Environment | Measured at 16 to 30 months of age
  StimQ READ Scale: Reading activity will be measured by using the StimQ Reading Scale. The StimQ is a structured interview. Individual items are summed, and scores range ranges from 0 to 19. Higher scores reflect higher reading activities.
Measurement of the Child's Home Environment | Measured at 16 to 30 months of age
  StimQ Parental Involvement in the Developmental Advance scale (PIDA). The prenatal involvement in child development will be measured by using the StimQ PIDA scale. The StimQ is a structured interview. Individual items are summed, and scores range ranges from 0 to 10. Higher scores reflect higher parent involvement.
Measurement of the Child's Home Environment | Measured at 16 to 30 months of age
  StimQ Parental Verbal Responsivity Scale (PVR). Parent verbal responsiveness will be measured using the StimQ Parental Verbal Responsivity Scale. The StimQ is a structured interview. Individual items are summed, and scores range ranges from 0 to 4. Higher scores reflect higher parent verbal responsiveness.
Parent beliefs questionnaire | Measured at 16 to 30 months of age
  Adult-child interaction quality assessment. The questioner elicits parental beliefs about the importance of language environment for language development and parental self-efficacy.
Language Development Snapshot (LDS) report | Measured at 16 to 30 months of age
  The Language Developmental Snapshot is a parent report that provides an estimate of child's developmental age with respect to receptive and expressive language skills.
Fidelity of implementation | Through study completion, an average of 1 year
  At each of the 10 LENA program sessions, a member of the Rice research team will attend (either virtually or in person) and collect data about Fidelity of Implementation of the LENA program, including liaison adherence to the material in the session, parental behavior at the session, liaison workload and preparation, as well as other measures of fidelity.
MacArthur Bates Communicative Development Inventories (CDI) | Measured at 16 to 30 months of age
  Parent questionnaire of receptive and expressive language skills. The inventory will be used to capture important information about children's developing abilities in early language. The Words and Sentences version is are appropriate for children 16-30 months. It contains a 100-word productive vocabulary checklist and a question about combining words. Standard scores are based on percentiles for age and sex and range from <1 to 99th percentile. Raw scores range from 0 to 680. Both higher standard scores and raw scores indicate better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Snejana Nihtaianova, PhD, Study Director — William Marsh Rice University
Locations (1):
- Alief ISD, Houston, Texas, United States